CLINICAL TRIAL: NCT02608008
Title: Safety and Efficacy of EchoNavigator System Release II (Philips, Andover, MA) During Structural Heart Interventions
Brief Title: Safety and Efficacy of EchoNavigator System Release II During Structural Heart Interventions
Acronym: EchoNav
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, PD Dr. med. Tobias Zeus, Heinrich-Heine University, Duesseldorf
Other Study IDs: EchoNav
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Imaging Techniques
Keywords: 3D-Ultrasound; Live X-rays; EchoNavigator System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Data analysis transfemoral aortic valve implantation: Periinterventional data analysis during structural heart procedures like transfemoral aortic valve implantation with and without the use of EchoNavigator System Release II.
  Interventions: Device: Data analysis
- Data analysis MitraClip: Periinterventional data analysis during structural heart procedures like MitraClip Implantations with and without the use of EchoNavigator System Release II.
  Interventions: Device: Data analysis
- Data analysis PFO: Periinterventional data analysis during structural heart procedures like PFO implantations with and without the use of EchoNavigator System Release II.
  Interventions: Device: Data analysis
- Data analysis ASD: Periinterventional data analysis during structural heart procedures like ASD implantations with and without the use of EchoNavigator System Release II.
  Interventions: Device: Data analysis

INTERVENTIONS:
Device: Data analysis — data parameters Analysis

SUMMARY:
The purpose of this study is to collect data regarding the safety and efficacy of EchoNavigator System Release II during structural heart interventions in the clinical practice. Data of procedures with and without the use of EchoNavigator System Release II will be collected, analysed and evaluated.

DETAILED DESCRIPTION:
EchoNavigator System Release II is a CE certified innovative periinterventional imaging modality used in our clinic of cardiology, pulmonology and angiology during structural heart interventions like transfemoral aortic valve Implantation (TAVI), MitraClip implantation, patent foramen ovale (PFO), atrial septal defect (ASD) and left atrial appendage (LAA). During this interventions EchoNavigator is able to combine live X-ray Images and 3D Echo guidance to enhance the efficiency of the procedure.

Specific periprocedural data parameter, e.g. procedure duration, radiation time, radiation dose, transseptal punction time (e.g.LAA) and contrast agent amount will be collected and analysed. The same data characteristics from the same procedures but without the periinterventional use of the EchoNavigator System Release II will be collected, analysed and compared with the data described above. A retrospective data collection between 2013 - 2017 of n=500 patients will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients of any ethnic origin aged > 18 years
* Signed and dated informed consent for the prospective study part

Exclusion Criteria:

* < 18 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients undergoing structural heart interventions like transfemoral aortic valve Implantation (TAVI), MitraClip implantation, patent foramen ovale (PFO), atrial septal defect (ASD) and left atrial appendage (LAA) with or without the periintervention use of the EchoNavigator System Release II.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-12-31 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of procedure time | baseline
  During interventions with and without the use of EchoNavigator System Release II

SECONDARY OUTCOMES:
Comparison of area dose product | baseline
  During procedures with and without the use of EchoNavigator System Release II
Comparison of contrast agent amount | baseline
  During procedures with and without the use of EchoNavigator System Release II
Comparison of data measurements of fluoroscopy time | baseline
  During procedures with and without the use of EchoNavigator System Release II
Comparison of duration of the transeptal punction | baseline
  During mitraClip implantations, ASD/PFO with and without the use of EchoNavigator System Release II.

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany